CLINICAL TRIAL: NCT04230187
Title: Bevacizumab Plus MFOLFOXIRI or MFOLFOX-6 As First-line Treatment for Patients with Unresectable Metastatic Colorectal Cancer: a Randomised, Open-label, Phase 3 Trial
Brief Title: Bevacizumab Plus MFOLFOXIRI As First-line Treatment for Patients with Unresectable Metastatic Colorectal Cancer
Acronym: TRIBE-C
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-18
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFOXIRI Plus Bevacizumab (Experimental): Patients will receive mFOLFOXIRI plus bevacizumab once every two weeks for 8 cycles as the first-line treatment.
  Interventions: Drug: mFOLFOXIRI plus Bevacizumab
- mFOLFOX6 Plus Bevacizumab (Active Comparator): Patients will receive mFOLFOX6 plus bevacizumab once every two weeks for 8 cycles as the first-line treatment.
  Interventions: Drug: mFOLFOX6 Plus Bevacizumab

INTERVENTIONS:
Drug: mFOLFOXIRI plus Bevacizumab — Bevacizumab (5 mg/kg on day 1) plus mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 8 cycles and followed by bevacizumab and fluoropyrimidine based maintence treatment
  Other Names: Oxaliplatin; Irinotecan; 5-Fluorouracil; Leucovorin; Bevacizumab
  Arms: mFOLFOXIRI Plus Bevacizumab
Drug: mFOLFOX6 Plus Bevacizumab — mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 8 cycles and followed by bevacizumab and fluoropyrimidine based maintence treatment
  Other Names: Oxaliplatin; 5-Fluorouracil; Leucovorin; Bevacizumab
  Arms: mFOLFOX6 Plus Bevacizumab

SUMMARY:
The current clinical trials and data on the triplet regimen combined with bevacizumab for first-line treatment of metastatic colorectal cancer were from European and American populations. The triplet regimens recommended by the NCCN and ESMO guidelines using irinotecan and 5-FU at a higher dose intensity cause a high incidence of adverse events in Asian population, and there was no high-quality data on efficacy in Chinese population, both of which have limited the clinical applications of the regimens in China. This study intends to conduct an improved triplet regimen (mFOLFOXIRI) combined with bevacizumab versus mFOLFOX6 combined with bevacizumab as a first-line multicenter, randomized, controlled phase III clinical trial in patients with advanced colorectal cancer. Progression-free survival (PFS), observable response rate (ORR), overall survival (OS), disease control rate (DCR), surgical resection rate, and safety and health-related quality of life (HRQoL) were assessed in the two groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

- Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.

Subjects with metastatic colorectal cancer(CRC) (Stage IV). Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 12 months of completion of adjuvant therapy.

Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study.

Metastatic CRC subjects must have measurable or non measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.

Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1. Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

- Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.

Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.

Heart failure grade III/IV (NYHA-classification). Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.

Subjects with known allergy to the study drugs or to any of its excipients. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.

Breast- feeding or pregnant women Lack of effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR).
Overall Survival (OS) | 5 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Toxicity assessed using the NCI common toxicity criteria, version 5.0. | 2 years
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No